CLINICAL TRIAL: NCT03988595
Title: Phase 1 Trial of Exercise Treatment With Concurrent First-Line Therapy for Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Exercise Treatment With Standard Therapy for Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-113
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hormone Receptor Positive Metastatic Breast Cancer
Keywords: Exercise; 19-113
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Exercise therapy will consist of individualized walking delivered 3 to 5 times weekly for 24 weeks. This trial will evaluate four escalated doses of exercise (90 mins/wk, 150 mins/wk, 225 mins/wk, 300 mins/week, or 375 mins/week).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- aerobic training 90 mins/wk (Experimental): Exercise sessions will consist of individualized, walking delivered following a non-linear(i.e., exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.
  Interventions: Other: Exercise Treatment
- aerobic training 150 mins/wk (Experimental): Exercise sessions will consist of individualized, walking delivered following a non-linear(i.e., exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.
  Interventions: Other: Exercise Treatment
- aerobic training 225 mins/wk (Experimental): Exercise sessions will consist of individualized, walking delivered following a non-linear(i.e., exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.
  Interventions: Other: Exercise Treatment
- aerobic training 300 mins/week (Experimental): Exercise sessions will consist of individualized, walking delivered following a non-linear(i.e., exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.
  Interventions: Other: Exercise Treatment
- aerobic training 375 mins/week (Experimental): Exercise sessions will consist of individualized, walking delivered following a non-linear(i.e., exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.
  Interventions: Other: Exercise Treatment

INTERVENTIONS:
Other: Exercise Treatment — Exercise sessions will consist of individualized, walking delivered following a non-linear (i.e.,exercise intensity is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule up to 7 individual treatment sessions/wk for 6 months. Remote supervised exercise sessions will be implemented and monitored using TeleEx. General physical activity as well as exercise performed outside of the structured treatment sessions will be evaluated via continuous monitoring using MSK approved telemedicine / wireless technology.

SUMMARY:
This study will test any good and bad effects of aerobic exercise performed while you are receiving the usual first-line treatment for metastatic breast cancer. The researchers think that exercise helps delay the development of resistance to hormone therapy while slowing the growth of tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, HR-positive (ER and/or PR), HER2-negative metastatic breast cancer (MBC)
* Postmenopausal status defined by lack of menses for 2 years, oophorectomy, or medical ovarian suppression
* Receiving first line endocrine-based therapy (tamoxifen, aromatase inhibitor, or fulvestrant; concurrent molecular therapy also allowed)
* Sedentary (i.e., <60 minutes / week of exercise)
* Age >18 years
* BMI ≥ 18.5
* Cleared for exercise participation as per screening clearance via PAR-Q+
* Cleared for study participation as per screening consultation with an MSK Exercise Physiologist
* Willingness to comply with all study-related procedures
* Patients with "treated and stable" brain lesions of a duration of ≥ 2 months may be enrolled

Exclusion Criteria:

* Life expectancy <6 months
* Enrollment onto any other therapeutic investigational study
* Mental impairment leading to inability to cooperate
* Concurrent participation in weight loss or other exercise programs

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 54 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
maximum feasible dose (MFD) | 24 weeks
  Feasibility is defined in terms of the relative dose intensive (RDI), the proportion of the planned exercise prescription that was completed without requiring a dose modification or interruption. The MFD is defined as the dose estimated to result in approximately 70% of patients achieving an RDI ≥ 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Indiana University (Data Collection Only), Indianapolis, Indiana
  - Johns Hopkins Hospital (Data Collection Only), Baltimore, Maryland
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Health Systems (Montefiore Medical Center) (Data Collection Only), The Bronx, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03988595/ICF_000.pdf